CLINICAL TRIAL: NCT04904692
Title: Virological and Immunological Monitoring in Patients (suspected Of/confirmed With) COVID-19
Acronym: Co-Vim
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); Chan Zuckerberg Initiative (Other); Flanders Institute for Biotechnology (Unknown)
Responsible Party: Sponsor
Other Study IDs: BC-07492
Record Dates: First submitted 2020-05-28; First posted 2021-05-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection; Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (plasma, PBMC), bronchoalveolar lavage fluid, nasopharyngeal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COVID-19 positive: Peripheral blood draw:
  * Day 1 of admission: blood draw.
  * Day 7-10 of hospitalization: blood draw.
  * Follow-up consultation: blood draw (selected patients).
  Bronchoscopic sampling:
  Material from bronchoscopic sampling (lavage fluid) will be collected only in those subjects in whom there is a diagnostic or therapeutic need for this procedure.
  Swabs for SARS-CoV-2 PCR:
  * Day 1 of admission: Extra oropharyngeal, nasal and nasopharyngeal (NP) swabs will be collected after the result of the initial diagnostic swab is known. In case of shortage of swabs, sputum samples will be collected as an alternative.
  * Day 7-14 of hospitalization: NP swab or clinically available alternative will be executed on day 7 repeated weekly.
  Interventions: Procedure: Blood draw; Procedure: Bronchoalveolar lavage; Procedure: SARS CoV-2 swabs
- COVID-19 negative: Peripheral blood draw:
  * Day 1 of admission: blood draw.
  * Follow-up consultation: blood draw (selected patients).
  Bronchoscopic sampling:
  Material from bronchoscopic sampling (lavage fluid) will be collected only in those subjects in whom there is a diagnostic or therapeutic need for this procedure.
  Swabs for SARS-CoV-2 PCR:
  o Day 1 of admission: Extra oropharyngeal, nasal and nasopharyngeal (NP) swabs will be collected after the result of the initial diagnostic swab is known. In case of shortage of swabs, sputum samples will be collected as an alternative.
  Interventions: Procedure: Blood draw; Procedure: Bronchoalveolar lavage; Procedure: SARS CoV-2 swabs

INTERVENTIONS:
Procedure: Blood draw — 8x9mL EDTA tubes. In subjects treated with hydroxychloroquine treatment an extra EDTA tube (4mL) will be collected for the REVIVE substudy.
Procedure: Bronchoalveolar lavage — Only in case of diagnostic or therapeutic indication.
Procedure: SARS CoV-2 swabs — Nasopharyngeal, oropharyngeal and nasal swabs

SUMMARY:
This study is a prospective, observational multicentric study. The study population entails adult patients hospitalized with a high clinical suspicion of COVID-19 and consists of two study arms (SARS-CoV2- vs. SARS-CoV2+).This combined fundamental research project has a dual goal: on the one hand assessing immunological predisposing factors for severe infection and investigating the immunological impact of SARS-CoV2 infection, on the other hand studying viral characteristics. Furthermore, a substudy will examine the pharmacokinetics and pharmacodynamics of hydroxychloroquine in patients receiving this antiviral treatment (REVIVE susbstudy). To answer these research questions, samples will be collected from patients with a high clinical suspicion of COVID-19, hospitalized at UZ Gent and 2 participating hospitals in Ghent (AZ Maria Middelares en AZ Jan Palfijn).

ELIGIBILITY:
Inclusion Criteria:

* Upper or lower respiratory symptoms and temperature ≥37.5°C, with high clinical suspicion of COVID-19
* Requiring hospitalization

Exclusion Criteria:

* Known pregnancy at the time of screening
* Inability to give informed consent or absence of legal representative who can give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients hospitalised with symptoms with upper or lower respiratory symptoms and temperature ≥37.5°C, with high clinical suspicion of COVID-19, who require hospitalisation.
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Identification of cytokines and chemokines associated with COVID-19 severity and outcome. | 6 months
  Cytokine and chemokine analysis (U-plex Mesoscale Diagnostics) on the plasma and BAL fluid will be correlated to disease severity and outcome
Identification of cellular subsets that can predict COVID-19 severity and outcome. | 6 months
  By using high-dimensional flow cytometry on cryopreserved PBMCs, the investigators will assess whether the phenotype and intracellular signaling can predict COVID-19 severity and disease outcome.
SARS CoV-2 sequencing. | 6 months
  Whole genome sequencing and viral metagenomics analysis will be performed on selected nasopharyngeal swabs and bronchoalveolar lavage fluid.

SECONDARY OUTCOMES:
Single-cell RNA sequencing of BAL fluid and matched PBMC samples. | 6 months
  Single -cell RNA sequencing will be performed on fresh BAL fluid and matched PBMCs by using 10X Genomics technology. The aim of the project is to study the transcriptional activity in different immune cells in the lung in COVID-19 patients with differing disease severity and compare these to non-COVID-19 respiratory infections.
Measurement of plasma hydroxychloroquine and N-desethylhydroxychloroquine (REVIVE). | 6 months
  In this pilot substudy (REVIVE study), the investigators aim to measure plasma hydroxychloroquine, measuring range 10-2250 ng/mL, and the active metabolite, plasma N-desethylhydroxychloroquine, measuring range 2-2250 ng/m, in patients treated with hydroxychloroquine.
Analysis of micronutrients Cu, Fe and Zn in plasma samples from COVID-19 + and COVID-19 - patients. | 12 months
  Total serum or plasma concentrations (mg/L) of Cu, Fe and Zn will be measured using a benchtop TXRF spectrometer (S4 T-STAR, Bruker Nano GmbH, Berlin, Germany) by prof. Gijs Du Laing and the laboratory of Prof. Lutz Schomburg.
Analysis of micronutrient Se in plasma samples from COVID-19 + and COVID-19 - patients. | 12 months
  Total serum or plasma concentrations (µg/L) of Se will be measured using a benchtop TXRF spectrometer (S4 T-STAR, Bruker Nano GmbH, Berlin, Germany) by prof. Gijs Du Laing and the laboratory of Prof. Lutz Schomburg.

CONTACTS AND LOCATIONS:
Overall Officials: Linos Vandekerckhove, Prof. MD, Principal Investigator — University Hospital, Ghent
Locations (3):
- Belgium (3):
  - AZ Jan Palfijn, Ghent, Oost-Vlaanderen
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - UZ Gent, Ghent, Oost-Vlaanderen

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 6 months